CLINICAL TRIAL: NCT06571929
Title: Effect of Task-Specific Training in Augmented Reality Context (INTERACT Protocol) on Upper Limb Function and Activities in Children With Spastic Cerebral Palsy: A Randomized Controlled Trial
Brief Title: Effect of Task-Specific Training in an Augmented Reality Context on Upper Limb Function and Activities in Children With Spastic Cerebral Palsy
Acronym: INTERACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Responsible Party: Principal Investigator, Luana Pereira Oliveira Gonçalves, Phd student, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Interventional
Record Dates: First submitted 2024-07-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral Palsy; Children; Games; Augmented reality
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Group control and experimental group
Who Masked: Outcomes Assessor
Masking Description: The study will be single-blind, meaning that the evaluator will not know the group to which the participant is assigned. Additionally, in the statistical analysis, the examiner will also remain blind regarding the type of intervention, referring to them as intervention 1 and intervention 2. However, the participants will not be blind to the treatments, due to the impossibility of blinding the type of intervention they will receive.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group INTERACT (Experimental): The INTERACT group will participate in an intervention with augmented reality games. During the games, participants will perform hand and arm movements, as well as activities such as sitting and standing up from a chair or climbing and descending steps. The augmented reality software to be used, BRAINN_XR, includes games such as puzzles and ping pong. The intervention will be conducted by physiotherapists trained in the use of the software. The sessions will take place three times a week, lasting 1 hour and 20 minutes, over a total period of 4 weeks.
  Interventions: Other: INTERACT
- Control group (No Intervention)

INTERVENTIONS:
Other: INTERACT — INTERACT is an individualized, task-specific training program that includes environmental enrichment, natural and augmented realities, and active training.
  Arms: Group INTERACT

SUMMARY:
Children with Cerebral Palsy (CP), a condition that affects movement and coordination, face difficulties in daily activities such as dressing, reaching for objects in high places, and getting up from seats. These challenges can negatively impact the quality of life for these children. Therefore, it is essential to seek effective treatments that help improve these skills.

The use of technology in treatments, especially with games that utilize augmented reality (AR), has proven to be a good strategy. This technique aids motor learning, improving the skills that children struggle with while also increasing motivation, allowing them to engage in activities they enjoy. However, the application of AR in children with CP is still limited.

In this context, it is crucial to provide appropriate treatments for these children, harnessing the benefits of AR technology. This study aims to investigate the effects of a protocol called "INTERACT protocol," which consists of training activities that interest children, such as reaching for objects and getting up from a bench. These activities are linked to AR games and will be conducted with accessible equipment for children with CP, aiming to improve their quality of life.

The children selected for the research will be divided into two groups: the experimental group (INTERACT) and the control group. This division will be done by random draw. The children in the control group will continue receiving the physiotherapy they are already undergoing for the same duration as the children in the INTERACT group. All children will participate in the treatment for 4 weeks, three times a week, with sessions lasting 1 hour and 20 minutes each.

Our hypothesis is that the children participating in the INTERACT protocol will show improvements in activities involving reaching for objects and in the transition from sitting to standing.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is defined as a group of permanent disorders of movement and posture development, caused by non-progressive brain injuries to the fetal or developing brain. The prevalence is 2.3 to 3.7 per thousand children born in low- and middle-income countries, and 1.6 to 2.9 per thousand children in developed countries.

The motor impairments present in children with CP are considered more complex in the upper limbs and are represented by changes in proprioception, selective motor control, presence of spasticity, reduced range of joint motion, muscle strength, and motor coordination deficits. These cited structural and functional impairments lead to limitations in the execution of activities, such as reaching and grasping, object manipulation, and activities of daily living.

Knowing that children with CP present deficiencies in upper limb motor function, it is important to carry out appropriate interventions. In this case, physiotherapy plays an important role in the rehabilitation of children with CP, but it is necessary to implement highly recommended approaches. The literature points to the level of evidence for improving motor function and task performance in children and adolescents with CP, highlighting specific task training, which is indicated with a green signal of scientific evidence and strong strength of recommendation.

Thus, rehabilitation for the recovery of function and motor activities involving the upper limbs of children with CP should focus on the practice of specific tasks used in daily life and real environments that are goal-directed. However, recent recommendations indicate that auxiliary interventions, when combined with specific task training, present better results. A new form of intervention that is expanding technology for rehabilitation and can be associated with specific task training is augmented reality (AR) therapy. AR has become an effective intervention strategy because it promotes motivation and interaction between the real world and the digital content universe, where both complement each other. It has been reported that AR training improves motor skills and provides the opportunity for low-cost rehabilitation, which can also be carried out at home. However, it is important to highlight that studies on AR are scarce and reveal gaps in the literature that need to be filled.

Given the need to fill these gaps, the objective of this study is to verify the effects of a specific task training protocol associated with augmented reality (INTERACT protocol) on the function and activities of the upper limbs in children diagnosed with spastic cerebral palsy.

Thus, the study will contribute new evidence for functional training in children with CP. The term INTERACT is derived from the English acronym, being a protocol of individualized exercises (I - individualized); task-specific (T - task-specific); with environmental enrichment (E - environment enrichment); utilizing augmented and real realities (RA - real and augmented realities); and conducted actively (act - active training). The INTERACT protocol will follow the principles of motor learning, and will be carried out with a low-cost AR equipment developed for rehabilitation, and a proposal for environmental enrichment with the insertion of real and virtual objects in the therapeutic environment.

Specific objectives:

To compare the effects of the INTERACT protocol with conventional physiotherapy treatment in children with spastic CP:

1. On the spatio-temporal and angular parameters of manual reach movement;
2. On recreational activities involving the upper limbs (UL);
3. On the transfer of learning, through the gain in performance of daily activities involving the upper limbs;
4. On motor learning retention, after a two-month follow-up period without intervention;
5. On postural sway during the sit-to-stand movement (with and without dual motor tasks) and during functional reach in standing.

Hypotheses:

It is expected that participants in the INTERACT protocol group will:

1. Improve spatio-temporal and angular parameters of manual reach movement, indicating better motor control;
2. Improve in recreational activities involving the upper limbs;
3. Improve performance in activities involving the upper limbs (transfer of learning to daily activities);
4. Retain motor learning after two months post-training;
5. Reduce postural sway during sit-to-stand movement and with dual motor tasks and during functional reach in standing.

Sample calculation:

It was performed a priori using the G*Power software. The effect size was determined based on the data (DASH scale) obtained in the study by Malick et al. (2022a), where an AR intervention for upper limb activities was performed. Thus, for the sample calculation, an effect size of 1.03, a statistical power of 90%, a confidence interval of 85%, and a statistical significance of 5% were considered, in an independent measures t-test analysis. The sample calculation resulted in a total of 34 participants. To ensure a sufficient number of participants at the end of the study, the inclusion of 4 more participants was established, to account for an estimated attrition rate of approximately 10%. Thus, the allocation of 19 participants in each of the two groups was determined.

Participants:

The study will consist of children with a medical diagnosis of unilateral and bilateral spastic CP, with a GMFCS (Gross Motor Function Classification System) level I and II, of both sexes, and aged between 6 and 12 years.

Randomization:

Children will be randomly allocated to the two intervention groups using an electronic allocation system: www.sealedenvelope.com. The children will be allocated to the group by block randomization of 6, stratified by GMFCS and MACS levels.

General Procedures:

Each participant will be evaluated. First, the parents will be presented with the Informed Consent Form, formalizing their consent and the child's participation in the project. The children will also sign the Informed Assent Form, which explains, in a less complex way, the entire study procedure and the steps the child will go through, and the child must assent. Volunteers from both intervention groups will be invited to participate in the study through advertisements on social media, such as Facebook, Instagram, and radio, as well as physical therapy clinics that agree to publicize the research by distributing flyers. If there is interest from the children and their guardians, the clinic will provide the researchers' contact information, allowing interested parties to contact the researchers.

Intervention:

Both the conventional physiotherapy treatment and the experimental treatment (INTERACT protocol) will be conducted over a period of 4 weeks, 3 times a week, with 1 hour and 20 minutes of training per day, by physiotherapists experienced in neuropediatrics and trained in this protocol. It is important to emphasize that the choice of frequency of 3 training sessions per week is based on the training typically used in rehabilitation settings in Brazil, which is considered feasible for children and their families. This choice of frequency was also based on recommendations found in the literature, such as those by Bailes et al. (2008) and McCoy et al. (2020), recommending at least 2 sessions per week.

Treatment Protocols:

First, the goals will be selected. The PEDI-CAT instrument (daily activities and mobility domains) has images in the application manual that will be used for the selection and visualization of goals.

INTERACT Protocol:

The protocol will be executed using augmented reality games through augmented reality software called BRAINN_XR. The software uses an RGB camera, a tool with electronic components and sensors, capable of tracking the child's gestures and movements in real-time. The child will initially be at a distance of 1.8m to 2.5m from the RGB camera, with a height of 0.6m to 1.2m from the ground, to have their body tracked and interact with the game interface. The real image of the child is projected into the game, allowing the visualization of both the game and the child on the screen.

The software has different games, including the puzzle game. The game will be projected onto the wall using a projector, and depending on the child's distance from the game, for example, greater distance, the pieces will be farther and higher or lower, directing more complex body movements such as squatting, stepping on a step, lateral walking, and functional reach beyond the support base. This allows for variations in activities involving the whole body. The game also provides auditory feedback when each piece is fitted and the number of hits and "Congratulations" at the end of the game.

Game Steps:

First, the theme, or the playful part of the game, will be set according to the participant's preferences.

To start the game, the participant will choose which limb they would like to start playing with, right or left, and the researcher will choose the challenges of the number of pieces, location of the pieces, environmental enrichment by inserting real objects into the virtual game, such as steps, benches of different heights, puzzle pieces, among others.

An example of a game: a virtual puzzle that requires movements such as picking up a piece at the bottom of the screen and taking it to the fitting location at the top of the screen. While the participant interacts with the virtual environment, they can also explore their surroundings, performing different movements with the whole body, according to the game's demands.

Control Group Intervention:

This group will receive treatment from the physiotherapist responsible for the intervention clinic. The treatment will aim at strengthening, active stretching, and biomechanical alignment. The resources used will be those typically employed in physiotherapy clinics, such as Swiss balls, benches, dumbbells, wall bars, and rollers, etc. With the clinic's authorization, the participants' records will be monitored weekly to check the types of exercises they are performing. We will offer the INTERACT treatment to this group if it demonstrates greater efficiency regarding the assessed outcomes.

Data Analysis SPSS 17 software will be used. The main focus of the study is the comparison of outcomes between the groups at the beginning and at the end of the intervention.

An intention-to-treat analysis will be applied (including all participants, regardless of the percentage of adherence to the treatment). Descriptive analysis will be performed for continuous and discrete data (mean and standard deviation (SD)). Continuous and discrete data that do not follow a normal distribution, even after data transformation, will be analyzed using non-parametric methods.

A MANOVA will be applied to compare the means of the outcomes of the experimental and conventional treatments. In both groups, for each variable of interest, the delta of the change between the end and the beginning of the intervention (Final score - Initial score) will be calculated. The delta will be used in all comparison analyses. Intragroup changes across the three assessments will use repeated measures MANOVA. Tukey's post hoc test will be used (comparison between the assessment before treatment, after treatment, and retention (2 months after the end of treatment)). The level of statistical significance will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* In the experimental and control groups, children who have been medically diagnosed with cerebral palsy, either unilateral or bilateral, with spasticity classification, will be included.
* Participants must be classified at GMFCS levels I and II, meaning they are capable of walking independently.
* The MACS (Manual Ability Classification System) should be between levels I (manipulates objects easily), II (manipulates most objects with reduced quality and speed), and III (manipulates objects with difficulty).
* The modified Ashworth score should be between 0 and 2.
* Ability to understand verbal commands and good comprehension of the proposed games.

Exclusion Criteria:

* Children with dystonic tone classification (identified by the Hypertonia Assessment Tool (HAT)), athetoid, or ataxic.
* GMFCS levels III, IV, and V.
* MACS levels IV and V.
* Modified Ashworth score of 3 to 4.
* Undergoing orthopedic surgical procedures within the past year.
* Receiving chemical blocks within the last 6 months.
* Deformities (muscle shortening and/or loss of joint mobility in the upper limbs) that prevent or compromise the ability to reach the midline.
* Presence of visual and/or auditory sensory deficits not corrected with devices.
* Use of medications that may alter muscle strength or tone.
* Cardiovascular limitations of any intensity, such as excessive fatigue, low exercise tolerance.
* Children who have undergone other intensive therapies within the past 6 months.
* Children with cognitive impairment indicated by caregivers or perceived by researchers due to difficulties in understanding verbal commands and virtual reality games.
* Children who do not accept playing augmented reality games.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Kinematic assessment of manual reach | Initial assessment (two days before the intervention); final assesment (maximum five days after the intervention);retention phase assessment (two months after the end of the intervention).
  Data collection of reach movement will be conducted using the OpenCap software, which combines computer vision and musculoskeletal simulation to quantify human movement kinematics from videos captured using iPhones.
Disabilities of the Arm, Shoulder and Hand (DASH) | Initial assessment (two days before the intervention); final assesment (maximum five days after the intervention);retention phase assessment (two months after the end of the intervention).
  This questionnaire measures physical disability and symptoms in single or multiple upper limb disorders. The DASH requires that the participant answers the questions based on their perceived condition from the previous week. If the participant did not have the opportunity to perform any of the activities in the questionnaire, they are instructed to estimate which response would be the most accurate. It does not matter which hand or arm is used to perform the activity; the questions should be answered based on the ability, regardless of how the task is performed. Participants must respond by circling the answers from 1 to 5, where 1 = there was no difficulty and 5 = could not do it. The higher the score, the greater the motor inability to perform daily activities involving upper limbs.
Assessment of postural sway during the sit-to-stand movement and during functional reach in standing position | Initial assessment (two days before the intervention); final assesment (maximum five days after the intervention);retention phase assessment (two months after the end of the intervention).
  These analyses will be performed using the force platform. Sitting to standing analysis: the child will be positioned on a height-adjustable bench with the knees, ankles and hips at a 90º angle, the upper limbs crossed and supported on the chest and the feet on the force platform in a symmetrical manner. Functional reach: on the force platform, with the lower limbs aligned at hip width, and the child should reach as far as possible, moving the center of mass forward, without taking the feet off the platform and with the shoulders flexed at 90º.

SECONDARY OUTCOMES:
The Canadian Occupational Performance Measure (COPM) | Initial assessment (two days before the intervention); final assessment (maximum five days after the intervention)
  Identify individual goals, satisfaction and performance for the execution of the experimental treatment. Participants should rate satisfaction and performance on a scale from 0 to 10 in relation to the activities chosen by the child, with 0 = low satisfaction and low performance and 10 = very good performance and high satisfaction.
Goal Attainment Scaling (GAS) | Initial assessment (two days before the intervention); intermediate assessment (after two weeks of training);final assessment (maximum five days after the intervention).
  It is described as a measure of individualized change, defining a set of unique goals for each person. The scoring scale reflects specific goals at five levels of achievement, ranging from -2 to +2, with -2 being much less than the expected outcome and +2 being much greater than the expected outcome.
Pediatric Evaluation of Disability Inventory (PEDI - CAT) | Initial assessment (two days before the intervention); final assesment (maximum five days after the intervention);retention phase assessment (two months after the end of the intervention).
  This instrument assesses functional abilities in four domains: (1) Activities of Daily Living; (2) Mobility; (3) Social/Cognitive; and (4) Responsibility. In this study, the Mobility domain will be used, which relates to the individual's performance in moving through various environments. After its application, the continuous score of the mobility domain will be used, which represents the child's current position along the function continuum and is not related to age.
Challenge Test | Initial assessment (two days before the intervention); final assesment (maximum five days after the intervention);retention phase assessment (two months after the end of the intervention).
  The Challenge Test contains 25 items that assess gross motor function, related to speed, balance, and coordination.The total score is 112 points and can be defined as follows: scores from 0 to 2 refer to the ability to perform the task, while scores from 3 to 5 refer to the speed of the item, with a score of 4 being given when the individual performs the task in the best possible way.
Dimensions of Mastery Questionnaire (DMQ) | Initial assessment (two days before the intervention); final assesment (maximum five days after the intervention);retention phase assessment (two months after the end of the intervention).
  This questionnaire contains six subscales: 1) object-oriented persistence; 2) gross motor persistence; 3) social persistence with adults and peers; 4) negative reactions to failure; 5) pleasure in mastery and general competence; 6) instrumental and expressive mastery motivation.There are 45 items scored on a 5-point scale ranging from 1 = not at all like this child to 5 = exactly like this child. The total motivation score will be considered before and after 4 weeks of treatment. The higher the scores, the greater the motivation.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Carlos (UFSCar), São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The primary and secondary outcome measures will be shared through publications in scientific journals.
Supporting Information: Study Protocol, CSR
Time Frame: The data will only be available once accepted for publication. The articles will be submitted for journal review at the end of 2024

REFERENCES:
- [Background] McIntyre S, Goldsmith S, Webb A, Ehlinger V, Hollung SJ, McConnell K, Arnaud C, Smithers-Sheedy H, Oskoui M, Khandaker G, Himmelmann K; Global CP Prevalence Group*. Global prevalence of cerebral palsy: A systematic analysis. Dev Med Child Neurol. 2022 Dec;64(12):1494-1506. doi: 10.1111/dmcn.15346. Epub 2022 Aug 11. PMID 35952356
- [Background] Alrashidi M, Wadey CA, Tomlinson RJ, Buckingham G, Williams CA. The efficacy of virtual reality interventions compared with conventional physiotherapy in improving the upper limb motor function of children with cerebral palsy: a systematic review of randomised controlled trials. Disabil Rehabil. 2023 Jun;45(11):1773-1783. doi: 10.1080/09638288.2022.2071484. Epub 2022 May 16. PMID 35575755
- [Background] Malick WH, Butt R, Awan WA, Ashfaq M, Mahmood Q. Effects of Augmented Reality Interventions on the Function of Upper Extremity and Balance in Children With Spastic Hemiplegic Cerebral Palsy: A Randomized Clinical Trial. Front Neurol. 2022 Jun 21;13:895055. doi: 10.3389/fneur.2022.895055. eCollection 2022. PMID 35800080
- [Background] Malick WH, Butt R, Awan WA, Ashfaq M, Mahmood Q. Effects of Augmented Reality Intervention on the Range of Motion and Muscle Strength of Upper Extremity in Children with Spastic Hemiplegic Cerebral Palsy: A Randomized Clinical Trial. Games Health J. 2022 Jun;11(3):168-176. doi: 10.1089/g4h.2021.0128. Epub 2022 Mar 14. PMID 35285674
- [Background] Jackman M, Sakzewski L, Morgan C, Boyd RN, Brennan SE, Langdon K, Toovey RAM, Greaves S, Thorley M, Novak I. Interventions to improve physical function for children and young people with cerebral palsy: international clinical practice guideline. Dev Med Child Neurol. 2022 May;64(5):536-549. doi: 10.1111/dmcn.15055. Epub 2021 Sep 21. PMID 34549424
- [Background] Novak I, Morgan C, Fahey M, Finch-Edmondson M, Galea C, Hines A, Langdon K, Namara MM, Paton MC, Popat H, Shore B, Khamis A, Stanton E, Finemore OP, Tricks A, Te Velde A, Dark L, Morton N, Badawi N. State of the Evidence Traffic Lights 2019: Systematic Review of Interventions for Preventing and Treating Children with Cerebral Palsy. Curr Neurol Neurosci Rep. 2020 Feb 21;20(2):3. doi: 10.1007/s11910-020-1022-z. PMID 32086598
- [Background] Levin MF, Demers M. Motor learning in neurological rehabilitation. Disabil Rehabil. 2021 Dec;43(24):3445-3453. doi: 10.1080/09638288.2020.1752317. Epub 2020 Apr 22. PMID 32320305